CLINICAL TRIAL: NCT01454427
Title: The Influence of Drugs Routinely Used in Cardiac Anesthesia on Impedance Aggregometry.
Brief Title: Influence of Anesthesia Drugs on Impedance Aggregometry
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Other Study IDs: 122/10
Record Dates: First submitted 2011-10-18; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Platelet Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy volunteers

SUMMARY:
Impedance aggregometry (IA) (Multiplate®)is a new whole blood platelet function test with potential use in anesthesia and intensive care. Most anesthetic drugs have been shown to have in vitro antiplatelet activity. The goal of this in vitro study is to evaluate the effect of several drugs, frequently used in cardiac anesthesia and intensive care, on platelet function as measured by IA

DETAILED DESCRIPTION:
Impedance aggregometry (IA) on the multiple platelet function analyzer (Multiplate®) ) is a whole blood point of care test evaluating platelet function. In IA, the increase in electrical impedance of whole blood is measured after the addition of a platelet activator. Some of the activators available are arachidonic acid (ASPI Test), ADP (ADP Test), TRAP-6 (TRAP Test) and collagen (COL TEST).

When an activator is added to the blood sample, the activated platelets will aggregate on the electrodes embedded in the test recipient. As platelets accumulate on the electrodes surface, the impedance will increase. The increase is measured and expressed in arbitrary units (AU). Reduced impedance implies platelet dysfunction or the presence of specific platelet inhibitors. For example, the ASPI test is inhibited in the presence of acetylsalicylic Acid and clopidrel inhibits the ADP test. Thrombin (TRAP) is an extremely potent agonist which can be used to monitor GpIIb/IIIa therapy.

The Multiplate® analyzer may have an important role in detecting and analyzing perioperative coagulopathies, but many drugs, routinely used in cardiac anesthesia or in the intensive care unit, have known in vitro antiplatelet effects, and may interfere with IA interpretation.

The goal of the study is to evaluate the influence of lidocaine, propofol, midazolam, and magnesium on the results of impedance aggregometry and to understand to which extent the tests are modified by the presence of one of these drugs.

20 healthy volunteers aged 18 to 65 years old will be recruited. Exclusion criteria are the use of non-steroidal anti-inflammatory drugs for 2 weeks prior to donation and known coagulation disorders. Whole blood is taken from the antecubital vein. Platelet count is measured. Blood samples for Multiplate® analysis are drawn in hirudin anticoagulated tubes. During storage, blood is gently moved in order to avoid sedimentation and spontaneous platelet aggregation.

For each sample baseline measurements are performed using ASPI Test, ADP Test, TRAP Test and COL Test.

The four study drugs are added to the blood samples, in isovolumic dilutions, to obtain subclinical, normal or near toxic plasma concentrations (table 1).

Study drugs low intermediate high Lidocaine (mcg/ml) 1 3 6 Magesium (mMol/l) 0.4 1 2.5 Midazolam (ng/ml) 150 250 500 Propofol (mcg/ml) 2 5 8 Table 1. Plasma concentration of the four study drugs

For every concentration, IA is measured using the 4 different activators. For every test and dose, the area under the curve is compared with the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old

Exclusion Criteria:

* Use of non-steroidal anti-inflammatory drugs for 2 weeks prior to donation.
* Known coagulation disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Drug induced platelet dysfunction as measured by impedance aggregometry.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo E Marcucci, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Morisoli AP, Gronchi F, Ferrari E, Blanc C, Frascarolo P, Angelillo-Scherrer A, Marcucci C. The influence of drugs used in cardiac anaesthesia and critical care on multiple electrode aggregometry: an in-vitro volunteer study. Eur J Anaesthesiol. 2014 Sep;31(9):499-504. doi: 10.1097/EJA.0000000000000113. PMID 25010745